CLINICAL TRIAL: NCT02974751
Title: Global Post-Market Registry Using Waterjet Ablation Therapy for Endoscopic Resection of Prostate Tissue
Acronym: OPEN WATER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Other Study IDs: TP0118
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: BPH
Keywords: Aquablation; AQUABEAM; BPH; LUTS
MeSH Terms: interventions — Aquablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Aquablation — Aquablation is a minimally invasive transurethral surgical procedure using the AQUABEAM system, a personalized image-guided waterject resection system that utilizes a high-velocity saline stream to resect and remove prostate tissue.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the AQUABEAM System for the treatment of Lower Urinary Tract Symptoms (LUTS) resulting from Benign Prostatic Hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Subject has diagnosis of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction or in urinary retention.
* Prostate size ≥ 20 mL and ≤ 150 mL as measure by TRUS.
* Patient is mentally capable and willing to sign a study-specific informed consent form.

Exclusion Criteria:

* Patients unable to stop anticoagulants, antiplatelet agents, or non-steroidal anti-inflammatory agents (NSAIDs, including aspirin greater or equal to 100mg) prior to treatment per standard of care.
* History of gross haematuria.
* Participants using systemic immune-suppressants including corticosteroids (except inhalants), known coagulopathy, or platelet disorder (except aspirin below 100mg/d).
* Contraindication to both general and spinal anesthesia.
* Any severe illness that would prevent complete study participation or confound study results.
* Subject is unwilling to accept a transfusion should one be required.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with lower urinary tract symptoms, including those with urinary retention, who meet all other enrollment criteria.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
IPSS score change | 3 months

CONTACTS AND LOCATIONS:
Locations (5):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia
- Asklepios Klinikum Harburg, Hamburg, Germany
- American University of Beirut Medical Center, Beirut, Lebanon
- Tauranga Urology Research, Tauranga, New Zealand
- Frimley Park Hospital, Frimley, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided